CLINICAL TRIAL: NCT06033053
Title: Real-time Neurofeedback Training of Fronto-limbic Areas Functional Connectivity to Reduce Arousal
Brief Title: Real-time Neurofeedback Training of Fronto-limbic Regions Functional Connectivity
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Electronic Science and Technology of China (Other)
Responsible Party: Principal Investigator, Benjamin Becker, Professor, University of Electronic Science and Technology of China
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: BAM_lab_MOST_05
Record Dates: First submitted 2023-08-28; First posted 2023-09-13 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Emotion Regulation; Healthy
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: Randomized active-sham group controlled between-subject: Group of healthy individuals will be randomly assigned to the experimental or the sham condition. The experimental group, will learn how to modulate the vmPFC-amygdala functional connectivity, while the sham group will try to modulate the functional connectivity of sham regions not involved in emotion regulation.
Who Masked: Participant, Investigator
Masking Description: The recruiter and the person in charge of conducting the experiment will be blind to the experimental condition, as will the participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group will learn how to modulate the vmPFC-amygdala functional connectivity while being presented with pictures inducing fear.
  Interventions: Device: Real-time fMRI neurofeedback from Turbo Brain voyager (TBV) 3.2
- Sham (Sham Comparator): The sham group will learn how to modulate the functional connectivity of sham ROIs while being presented with pictures inducing fear.
  Interventions: Device: Real-time fMRI neurofeedback from Turbo Brain voyager (TBV) 3.2

INTERVENTIONS:
Device: Real-time fMRI neurofeedback from Turbo Brain voyager (TBV) 3.2 — The two groups will undergo the same paradigm while learning to modulate the vmPFC -amygdala pathway and the sham pathway.

SUMMARY:
This is randomized active-sham group controlled between-subject real-time fMRI neurofeedback trial aimed at modulating the ventromedial prefrontal cortex (vmPFC)-amygdala pathway to control subjective anxiety and arousal.

DETAILED DESCRIPTION:
The present randomized active-sham group controlled between-subject real-time fMRI neurofeedback trial aims at determining if (1) subjects can gain volitional control over the vmPFC-amygdala pathway involved in implicit emotion regulation and arousal by means of connectivity informed neurofeedback, (2) whether the training has specific effects on the behavioral and psychophysiological arousal level, and (3) or the amygdala or the vmPFC connectivity, respectively.

The present project will determine the efficacy of the modulation of the vmPFC-amygdala functional connectivity pathway using vmPFC-amygdala upregulation (n = 25 subjects) compared to a sham control condition (targeting pathways not involved in emotion regulation, n = 20).

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old
* other genders
* No past or current psychiatric or neurological or other main disorders.

Exclusion Criteria:

* Pregnant, taking oral contraceptives
* Current use of medications
* Contraindication to MRI scanning (e.g., metal implants, claustrophobia or other conditions that make them inappropriate for MRI scanning).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Functional connectivity computed from blood oxygenation level dependent (BOLD) functional magnetic resonance imaging between regions of interest. | 40 minutes
  Increased functional connectivity computed from BOLD fMRI over the course of the real-time NF-fMRI training sessions in the neurofeedback group (regions of interest: bilateral amygdala and prefrontal area) but not in the sham group (regions of interest: bilateral motor cortex and primary auditory areas). Functional connectivity strength will be represented by bivariate regression coefficients from a general linear model characterizing the association between their BOLD signal timeseries

SECONDARY OUTCOMES:
Level of behavioural arousal assessed on NRS from 0 to 10 | 10 minutes
  After the presentation of movie clips inducing strong fearful emotions, the participant will rate the behavioural level of arousal on a Numeric Rating Scale (NRS) from 0 (lowest level of arousal) to 10 (highest level of arousal). The neurofeedback group will present lower level of arousal in comparison to the sham group.

OTHER OUTCOMES:
Level of behavioural anxiety assessed on NRS from 0 to 10 | 10 minutes
  After the presentation of movie clips inducing strong fearful emotions, the participant will rate the behavioural level of anxiety on a Numeric Rating Scale (NRS) from 0 (lowest level of anxiety) to 10 (highest level of anxiety). The neurofeedback group will present lower level of anxiety in comparison to the sham group.

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Becker, Ph.D., Principal Investigator — University of Electronic Science and Technology of China
Locations (1):
- University of Electronic Science and Technology of China, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No